CLINICAL TRIAL: NCT06076200
Title: Population Pharmacokinetic of Piperacillin/Tazobactam in Maternal and Neonatal Populations With High Risk for EOS
Brief Title: Population Pharmacokinetic of Piperacillin/Tazobactam in Maternal and Neonatal Populations
Status: Recruiting | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: SDU-2023-PPK-005
Record Dates: First submitted 2023-09-23; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Early-Onset Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Piperacillin; Tazobactam; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Biological samples include blood samples, amniotic fluid samples, placenta samples, maternal milk samples in pregnant women and umbilical cord blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Piperacillin Sodium and Tazobactam Sodium for Injection — Piperacillin/Tazobactam, specification: 4g; 0.5g. Anti-infective therapy with piperacillin/tazobactam, specific regimen based on clinical practice, without intervention.

SUMMARY:
The purpose of this study is to describe the population pharmacokinetic characteristics of piperacillin/tazobactam after intravenous administration in pregnant women during pregnancy and delivery, and to evaluate pharmacodynamic effectiveness and safety of piperacillin/tazobactam in pregnant women whose baby are at high risk of developing early-onset sepsis after birth.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old;
* Pregnant women whose baby are at high risk of developing early-onset sepsis after birth have indications to use preventive or therapeutic antibiotics, and the antibiotics used are PIP/TAZO；
* Patients and their families are fully aware of the research content and sign the informed consent form.

Exclusion Criteria:

* Intolerance or serious adverse reactions to antibiotic use;
* Patients who stopped using PIP/TAZO more than 24 hours before delivery;
* Receiving other systemic trial drugs;
* There are other factors that the researchers think are not suitable for inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research population of this study is pregnant individuals whose baby at high risk of developing early-onset sepsis after birth.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clearance (L/h) of piperacillin/tazobactam | Through study completion, an average of 20 days.
  The mean population pharmacokintic parameter as well as its interindividual variability
Volume of Distribution (L) of piperacillin/tazobactam | Through study completion, an average of 20 days.
  The mean population pharmacokintic parameter as well as its interindividual variability

SECONDARY OUTCOMES:
PD target attainment | Through study completion, an average of 20 days.
  PD target is defined as the time of free drug concentration beyond MIC during the dose interval
Adverse events | Through study completion, an average of 20 days.
  Drug-related adverse events and serious adverse events during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Principal Investigator — Shandong University
Locations (1):
- Shandong Provincial Hospital, Jinan, China

IPD SHARING:
Plan to Share IPD: Undecided